CLINICAL TRIAL: NCT04829461
Title: Clinical Investigation to Evaluate the Effectiveness of the Ambu® aScope™ 4 Cysto With the Ambu® aView™ 2 Advance for Flexible Cystoscopy
Brief Title: Effectiveness of Ambu® aScope™ 4 Cysto With the aView™ 2 Advance for Flexible Cystoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ambu Inc. (Industry)
Collaborators: Ambu A/S (Industry)
Responsible Party: Sponsor
Organization: Ambu A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIS-023
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Cystoscopy; Ureteral Stent
Keywords: Ureteral Stent; aScope 4 Cysto; single-use cystoscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Ambu® aScope™ 4 Cysto (Experimental): Ureteral stent removal procedure performed with Ambu® aScope™ 4 Cysto (single-use cystoscope).
  Interventions: Device: Ambu® aScope™ 4 Cysto with the aView™ 2 Advance used for stent removal
- Standard of Care (SOC) (Active Comparator): Ureteral stent removal procedure performed with standard of care (reusable cystoscope).
  Interventions: Device: Standard of care reusable cystoscope used for stent removal

INTERVENTIONS:
Device: Ambu® aScope™ 4 Cysto with the aView™ 2 Advance used for stent removal — Procedure using a single-use cystoscope for stent removal
  Arms: Ambu® aScope™ 4 Cysto
Device: Standard of care reusable cystoscope used for stent removal — Procedure using a reusable cystoscope for stent removal
  Arms: Standard of Care (SOC)

SUMMARY:
The purpose of this study is to evaluate the use of the single-use Ambu® aScope™ 4 Cysto for removal of ureteral stents as compared to routine flexible reusable cystoscopes.

DETAILED DESCRIPTION:
This study is a prospective, randomized, multi-center, post-market investigation of the effectiveness of Ambu® aScope™ 4 Cysto (single-use cystoscope) as compared to routine flexible reusable cystoscopes (standard of care) for ureteral stent removals. The investigation will include approximately 102 subjects (randomized at a 1:1 ratio).

ELIGIBILITY:
Inclusion Criteria:

1. Adult (male or female), ≥18 years old
2. Patient undergoing routine flexible cystoscopy
3. Patient with a ureteral stent in the urinary system that is ready to be removed.
4. No active urinary tract infection
5. Subject is willing and able to sign informed consent and HIPAA authorization and comply with requirements of the protocol.

Exclusion Criteria:

1. History of prior bladder/urethral reconstructive surgery.
2. History of high-grade bladder cancer or carcinoma in-situ of the bladder, undergoing cystoscopy for follow-up/surveillance purposes.
3. Known unpassable urethral stricture
4. Febrile patient with active urinary tract infection (UTI)
5. Subjects with acute infection (acute urethritis, acute prostatitis, acute epididymitis)
6. Subject with severe coagulopathy
7. Patient is unable to read and/or understand study requirements
8. Patient is unable or unwilling to provide written consent to participate in the study.
9. Subject, in the opinion of the Investigator, has a severe comorbidity, poor general physical/mental health and/or a condition that will not

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
The success rate of the Ambu® aScope™ 4 Cysto and the Ambu® aView™ 2 Advance for stent removal procedures performed in the outpatient setting. | Procedure Date (Day 0)
  Stent removal procedural success rate with the Ambu® aScope™ 4 Cysto and the Ambu® aView™ 2 Advance.

SECONDARY OUTCOMES:
Comparison of Ambu® aScope™ 4 Cysto and the Ambu® aView™ 2 Advance for stent removal procedures performed in the outpatient setting to standard of care reusable scopes on scope performance. | Procedure Date (Day 0)
  Comparison of Ambu® aScope™ 4 Cysto and the Ambu® aView™ 2 Advance for stent removal procedures performed in the outpatient setting to standard of care reusable scopes on scope performance as measured by procedure success rates, conversion rates, and device deficiency rates.
Comparison of the Cumulative Procedure Time between the Ambu® aScope™ 4 cysto and the site's SOC reusable flexible cystoscope. | Procedure Date (Day 0)
  Comparison of the Cumulative Procedure Time between the Ambu® aScope™ 4 cysto and the site's SOC reusable flexible cystoscope as measured by:
  1. Scope preparation for procedure
  2. Actual procedure time (insertion of cystoscope to removal of cystoscope) and
  3. Time to dispose of or prepare for reprocessing of cystoscopy equipment.
To evaluate the user experience during cystoscopic procedures. | Clinician Questionnaire; completed within one (1) day of procedure date (Day 0).
  Clinician satisfaction rated on a five-point scale (1-5) with 5 being the better outcome.
  1. Ease of insertion
  2. Ability to visualize anatomical landmarks and/or urothelium changes
  3. Perception of image quality
  4. Maneuverability in the bladder
  5. Scope articulation with tools in the working channel
  6. Visualization while tools are in the working channel
Safety Endpoints | 7-10 Days Post-Procedure
  Safety will be assessed based on the incidence rates of adverse events based on the seriousness and relatedness to the device and/or procedure.
  1. All reported device and/or procedural related adverse events through ten (10) days post-procedure
  2. All Serious Adverse Events (SAEs) through 10 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Smith, Study Director — Ambu Inc.
Locations (3):
- United States (3):
  - The Pennsylvania State University and The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samplaski MK, Jones JS. Two centuries of cystoscopy: the development of imaging, instrumentation and synergistic technologies. BJU Int. 2009 Jan;103(2):154-8. doi: 10.1111/j.1464-410X.2008.08244.x. Epub 2008 Dec 8. PMID 19076146
- [Background] O'Sullivan DC, Chilton CP. Flexible cystoscopy. Br J Hosp Med. 1994 Apr 6-19;51(7):340-5. PMID 8081563
- [Background] Pillai PL, Sooriakumaran P. Flexible cystoscopy: a revolution in urological practice. Br J Hosp Med (Lond). 2009 Oct;70(10):583-5. doi: 10.12968/hmed.2009.70.10.44626. PMID 19966704
- [Background] Gee JR, Waterman BJ, Jarrard DF, Hedican SP, Bruskewitz RC, Nakada SY. Flexible and rigid cystoscopy in women. JSLS. 2009 Apr-Jun;13(2):135-8. PMID 19660204
- [Background] Kadi N, Menezes P. ABC of flexible cystoscopy for junior trainee and general practitioner. Int J Gen Med. 2011;4:593-6. doi: 10.2147/IJGM.S20267. Epub 2011 Aug 19. PMID 21887113
- [Background] Miner N, Harris V, Lukomski N, Ebron T. Rinsability of orthophthalaldehyde from endoscopes. Diagn Ther Endosc. 2012;2012:853781. doi: 10.1155/2012/853781. Epub 2012 May 16. PMID 22665966
- [Background] Sokol WN. Nine episodes of anaphylaxis following cystoscopy caused by Cidex OPA (ortho-phthalaldehyde) high-level disinfectant in 4 patients after cytoscopy. J Allergy Clin Immunol. 2004 Aug;114(2):392-7. doi: 10.1016/j.jaci.2004.04.031. PMID 15316522
- [Derived] Johnson BA, Raman JD, Best SL, Lotan Y. Prospective Randomized Trial of Single-Use vs Reusable Cystoscope for Ureteral Stent Removal. J Endourol. 2023 Oct;37(10):1139-1144. doi: 10.1089/end.2023.0134. PMID 37565290